CLINICAL TRIAL: NCT05568732
Title: Comparative Evaluation of Treatment Outcome of Volume Stable Collagen Matrix in Isolated Labial rt2 Gingival Recession as Compared to Subepithelial Connective Tissue Graft : a Randomized Controlled Clinical Trial.
Brief Title: Evaluation of Volume Stable Collagen Matrix in RT2 Gingival Recession Compared to Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: vaishali pagade perio 22/29
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Scaling and root planing will be performed and after resolution of gingival inflammation, root coverage procedure will be done with VCMX using minimally invasive access technique.
  Interventions: Procedure: Root coverage procedure will be done with VCMX
- Control group (Active Comparator): Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with CTG using minimally invasive access technique.
  Interventions: Procedure: Root coverage procedure will be done with CTG

INTERVENTIONS:
Procedure: Root coverage procedure will be done with VCMX — Scaling and root planing will be performed and after resolution of gingival inflammation, root coverage procedure will be done with VCMX using minimally invasive access technique.
  Arms: Test group
Procedure: Root coverage procedure will be done with CTG — Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with CTG using minimally invasive access technique.
  Arms: Control group

SUMMARY:
Gingival recession is the migration of the gingiva to a point apical to the cemento-enamel junction. In order to treat challenging miller class 3 or RT2 recessions, several mucogingival approaches have been proposed. The subepithelial connective tissue graft (CTG) combined with a coronally advanced flap (CAF) has been considered as the "gold standard" for recession coverage around teeth. However, significant resorption of CT graft material has been reported if the graft material is exposed. And that can reduce the possibility of complete root coverage. volume stable collagen matrix - (VCMX ) is a volume stable, fully resorbable, porous, collagen matrix of porcine origin and spongious consistency and is one of the most biocompatible, novel material to be used in this study. VCMX of porcine origin is predominantly made of collagen type I and III and a small portion of elastin. VCMX is able to overcome the volume stability limitation of most commercially available grafts. The surgical technique proposed in a case series using a volume-stable collagen matrix and autogenous subepithelial CTG may be an effective method for periodontal biotype modification through thickening of the entire facial aspect for the treatment of gingival recession. VCMX consists of a single porous layer with interconnected pores (93% volume porosity) and an average pore size of 92 µm. While mechanical stability is achieved by chemical crosslinking, mechanical testing demonstrated preserved elasticity of the material over 14 days. Data have convincingly demonstrated enhanced promigratory and proadhesive properties of three primary cell types human oral fibroblas(hOFs) and human umblical vein endothelial cells(HUVECs), grown on the VCMX. The VCMX was characterized with an efﬁcient adsorption of four recombinant growth factors (TGF-β, PDGF-BB, FGF-2, and GDF-5), naturally present in the blood clot. And in a RCT with Miller's class 1 and 2 it also showed that it provides volume stability and withstands early resorption, while encouraging formation of new soft tissue. Due to its wettability, suture-ability and biological properties, the device has been reported to become well integrated with surrounding soft tissue. No study has been evident on comparing VCMX and SCTG for Miller's class 3/RT2 recession defect. Therefore the purpose of the study is to compare the clinical outcome of VCMX ans SCTG in Miller's class 3/RT2 .

DETAILED DESCRIPTION:
Gingival recession is the migration of the gingiva to a point apical to the cemento-enamel junction. In routine dental practice gingival recession defects are frequently encountered complain because of functional and esthetic concern of patients . Indications of root coverage procedures including esthetics, defect progression, hypersensitivity, or difficulties with oral hygiene support the use of periodontal plastic surgical procedures.

Miller in 1985 proposed a classification system which is probably the most commonly employed system to classify gingival recession and divided it into four categories. Class III recession extends to or beyond the MGJ with bone or soft tissue loss in the interdental area, or there is malpositioning of the teeth which may be a hinderance to complete root coverage and hence partial root coverage can be expected. According to Cairo (2011), Recession Type 2 (RT2): Gingival recession associated with loss of interproximal attachment. The amount of interproximal attachment loss (measured from the interproximal CEJ to the depth of the interproximal pocket) was less than or equal to the buccal attachment loss (measured from the buccal CEJ to the depth of the buccal pocket) .

The subepithelial connective tissue graft (CTG) combined with a coronally advanced flap (CAF) has been considered as the "gold standard" for recession coverage around teeth, Harvesting of SECTG can be done from the palate, maxillary tuberosity or edentulous ridges. The palate remains the most common donor site. The harvesting of SECTGs produces less postoperative morbidity than free gingival grafts. Many modifications of the techniques to harvest SECTGs have been proposed, each subtly different from each other in the number of incisions, flap design, and technique. Hurzeler suggested a single incision technique to harvest SECTG, with advantages of healing with primary intention at the donor site and very less postoperative morbidity to the patient but in the quest for easier to use, unlimited supply alternatives to painful harvest grafts, researchers continue to test harvest graft substitute. However, the harvesting procedure is classified as being difficult and may be associated with the risk of intra and postoperative complications such as bleeding, infection or necrosis. Several studies have focused on alternatives including human dermis and collagen matrices(CMX). A multicentre trial in isolated recessions indicated that the addition of CMX to coronally advanced flap resulted in a significant benefit in terms of marginal soft tissue thickness and patient-reported outcomes compared to coronally advanced flaps alone.The results, however, failed to support the non-inferiority hypothesis of CMX with respect to CTG in terms of root coverage. Now, a volume stable, fully resorbable, porous, collagen matrix of porcine origin and spongious consistency (volume stable collagen matrix - VCMX ) has become available for soft tissue augmentation. The surgical technique proposed in a case series using a volume-stable collagen matrix and autogenous subepithelial CTG may be an effective method for periodontal phenotype modification through thickening of the entire facial aspect for the treatment of gingival recession. In a Randomized clinical trial(RCT), it showed that VCMX provides volume stability and withstands early resorption, while encouraging formation of new soft tissue. Due to its wettability, suture ability and biological properties, the device has been reported to become well integrated with surrounding soft tissue.

Given these characteristics, this study will be conducted to evaluate the root coverage % in Miller's class 3 or RT2 gingival recession in mandibular anterior teeth using a VCMX compared to CTG with minimally invasive access technique.

The present randomized controlled clinical trial will be conducted in the department of Periodontics and Implantology, Post Graduate Institute of Dental Sciences, Rohtak. Study design is of 12-14 months. Patients will be recruited from the outpatient department of periodontology. It will be divided into Test group - VCMX Scaling and root planing will be performed and after resolution of gingival inflammation, root coverage procedure will be done with VCMX using minimally invasive access technique and Control group - CTG Scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage procedure will be done with CTG using minimally invasive access technique.

Full mouth scaling and root planing will be performed using ultrasonic and hand instruments as needed.

After administration of local anaesthesia, exposed root surface will be scaled and planned using curettes. With a minimally invasive access technique a full thickness tunnel will be prepared with the aid of specific tunnelling instruments, extending it sufficiently beyond the mucogingival line into alveolar mucosa. This will be done to completely releasing the tunnel-papillae complex, thus facilitating its passive coronal replacement.

CTG will be procured from the palate or tuberosity area for root coverage procedure by single incision technique. The template will be placed on the palate to mark the extent of the graft, after local anesthesia was administered. The palatal wound will be sutured to obtain primary wound closure. VCMX was thinned and cut to size for the defect, rounding and sloping the matrix edges so they were thinner around the perimeter. In test group, Volume-stable collagen matrix will be placed and in control group only CTG will be placed.

Suitable antibiotics and analgesics will be prescribed for 5 days. Chlorhexidine (0.12%) mouthwash will be advised till suture removal. The dressing and sutures will be removed after 7-10 days. Instructions will be given for gentle brushing with a soft toothbrush and reinstructed for proper oral hygiene maintenance.

The patient will be recalled for examination weekly for upto 1 month after surgery and again at 3, 6 and 9 months.

After enrollment, participants will be instructed about oral hygiene maintainance and undergo nonsurgical periodontal treatment in the form of scaling and root planing. All baseline parameters will be recorded 4-6 weeks after SRP after once gingival inflammation is resolved. Placement of VCMX will be done in the Test group and participants will be recalled after 3 months for recording all parameters. Among the control group participants, CTG will be placed after resolution of gingival inflammation ( 4-6 weeks after SRP ). Both groups will be re-evaluated and undergo recording of all parameters at the end of final treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with Millers class3[4] or RT2[6] isolated recession defects in labial mandibular anterior teeth region.
* 2. Systemically healthy individuals.
* 3. Absence of clinical tooth mobility.
* 4. Age 18-45 years old.
* 5. A full mouth plaque index < 20%
* 6. Patient showing adequate compliance and willing to participate in the study.

Exclusion Criteria:

* Patients having systemic disease such as hypertension, diabetes, hyperthyroidism or on medication that influence the outcome of periodontal therapy.
* Previous surgical attempt to correct gingival recession.
* Crowding of affected teeth.
* Patients with active periodontal disease.
* Smokers and tobacco users.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Root coverage percentage | 9 months
  Percentage of root coverage will be calculated by using pre and post operative recession depth

CONTACTS AND LOCATIONS:
Overall Officials: VAISHALI PAGADE, BDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Post Graduate Institute Of Dental Science, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No